CLINICAL TRIAL: NCT06749327
Title: Ultra-processed Foods, Diet Quality, and Cardiometabolic Health
Brief Title: Dissecting the Roles of High-quality Diets and Ultra Processed Foods on Cardiometabolic Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: University College Dublin (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Jayne Woodside, PhD, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TBC
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Cardiometabolic Risk Factors
Keywords: Plant-based diets; Diet quality; Cardiometabolic risk factors; Ultra-processed foods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High UPF, high hPDI diet (Experimental): High ultra-processed foods (UPFs) and healthy plant based diet
  Interventions: Behavioral: High UPF, high hPDI diet
- Low UPF, high hPDI diet (Active Comparator): Low ultra-processed foods (UPFs) and high healthy plant-based diet
  Interventions: Behavioral: Low UPF, high hPDI diet

INTERVENTIONS:
Behavioral: High UPF, high hPDI diet — High ultra-processed foods (UPFs) and healthy plant based diet
  Arms: High UPF, high hPDI diet
Behavioral: Low UPF, high hPDI diet — Low ultra-processed foods (UPFs) and high healthy plant-based diet
  Arms: Low UPF, high hPDI diet

SUMMARY:
Controversy remains around the role of ultra-processed food (UPF) consumption and health outcomes. A key question that remains to be answered is: when diet quality is the same, does food processing itself have any independent health effects? The current application aims to isolate the health effects of food processing from those of diet quality through the conduct of a dietary intervention study.

DETAILED DESCRIPTION:
Controversy remains around the role of UPF consumption and health outcomes. A key question that remains to be answered is: When diet quality is the same, does food processing itself have any independent health effects?

The current study aims to isolate the health effects of food processing from those of diet quality through the conduct of a dietary intervention study.

To isolate the health effects of food processing, the investigators propose to use healthy plant-based diets as the "base" diet. The investigators propose to initially discover plasma metabolomic features responsive to improved hPDI adherence and then conduct a dietary intervention trial to evaluate the impact of UPF consumption, in the setting of a high hPDI diet, on cardiometabolic outcomes and metabolic pathways.

The study will consist of a run-in phase where participants with a low adherence to a plant based diet will be randomized into (1) an intervention group that will receive diet counselling to follow a high hPDI diet over a period of 6 weeks and (2) a control group that will consume their usual diet (low hPDI). Both arms will be advised to avoid ultra processed food (UPF) consumption. Assuming 15% attrition, the study will enrol 118 participants for the run-in phase. Individuals with a high adherence to plant based diet will follow their normal diet for the 6 weeks of this run-in phase and then will be randomised into the main 4 month study.

In the main four month study, a randomized controlled parallel group dietary intervention will be conducted in participants with high hPDI in Ireland (North and South) to evaluate the impact of UPF consumption, in the context of a high hPDI diet, on cardiometabolic outcomes such as glycated haemoglobin and total cholesterol, and metabolic pathways. Participants will be randomized into one of 2 groups: high UPF hPDI diet or low UPF hPDI diet. Assuming an attrition rate of 15%, the study will enrol ~212 individuals to achieve a sample size of 180 participants who will complete the trial.

Randomization will be performed using a randomization scheme generated using www.randomization.com with random block sizes by research staff independent of the study. The investigators will stratify randomization according to age and BMI.

Power calculation : Assuming a change in total cholesterol of 9 mg/dL at four months and assuming a SD of change of 20, a total of 78 participants in each group is needed. Allowing for participant dropout of 15%, which is similar to that observed in the investigator's previous interventions, gives an overall sample size of 180.

Based on an SD of difference in change in HbA1c of 0.3%, the same sample size could detect as statistically significant a difference in HBA1c of 0.15% between the two intervention groups at four months.

The total number of participants that will be enrolled will be 330: 118 (run-in phase) and 212 (4 month trial).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 65 years in general good health with BMI < 35 kg/m2 who can provide informed consent.

Exclusion Criteria:

* Participants will be ineligible to enrol if they have diabetes, CVD, any type of cancer (except for basal cell skin cancer), or a condition (pregnancy, breastfeeding, etc) or dietary restriction(s) that would substantially limit their ability to complete the study.

Individuals will be screened for their adherence to the Plant based diet Index (PDI ).

1. Individuals with low adherence will enter run-in phase only (6 weeks)
2. Individuals with high adherence will enter the main intervention (4 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1C) (mmol/mol) | Baseline and 4 months
  Change in HbA1c over the course of the 4 month intervention.
Total cholesterol (mg/dL) | Baseline and 4 months
  Change in total cholesterol will be measured over the course of the 4 month intervention.

SECONDARY OUTCOMES:
Anthropometric measure: Weight (kg) | Baseline and 4 months
  Weight (kg) measured using calibrated scales at baseline and 4 months
Anthropometric measure: Height (m) | Baseline and 4 months
  Height (m) measured using stadiometer at baseline and 4 months.
Anthropometric measure: Waist circumference (cm) | Baseline and 4 months
  Waist circumference (cm) measured at baseline and 4 months.
Anthropometric measure: Hip circumference (cm) | Baseline and 4 months
  Hip circumference (cm) measured at baseline and 4 months.
Blood pressure (mmHg) | Baseline and 4 months
  Blood pressure will be measured twice from the right arm, using an automated Omron sphygmomanometer, with the participant sitting quietly for at least five minutes in advance
Dietary assessment | Baseline and 4 months
  2x 24-hour dietary recalls
Physical activity | Baseline and 4 months
  Questionnaire/objective physical activity monitor. Higher scores in both questionnaire and physical activity monitor will indicate improved outcome.
Demographic/lifestyle information | Baseline and 4 months
  E.g. alcohol use, medication use.
Continuous Glucose Monitoring (mmol/L) | Baseline and 4 months
  Continuous glucose monitoring (mmol/L) at baseline and 4 months
Plasma metabolome | Pre and post run-in phase (6 week run-in) ; baseline and 4 months (main trial)
  Fasting blood samples will be drawn from the antecubital vein and immediately separated into plasma.
Gut microbiome | Baseline and 4 months
  Stool samples will be collected at home within 24 h of the study visit and brought to the laboratory for storage. Samples will be profiled for gut microbiota composition and functional potentials.
Inflammatory markers e.g. CRP (mg/L) | Baseline and 4 months
  Changes in inflammatory markers such as CRP (mg/L) over the course of the 4 month intervention

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Lorraine Brennan, PhD, Principal Investigator — University College Dublin
Locations (2):
- University College Dublin, Dublin, Ireland, Ireland
- Centre for Public Health, Queen's University Belfast, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided